CLINICAL TRIAL: NCT03768297
Title: Clinical Evaluation of Soft Tissue Esthetics Around Immediate Implant Using Dual Zone Therapeutic Concept Versus Buccal Gap Fill to Bone Level.A Randomized Controlled Clinical Trial
Brief Title: Clinical Evaluation of Soft Tissue Esthetics Around Immediate Implant Using Dual Zone Therapeutic Concept Versus Buccal Gap Fill to Bone Level
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, RWGWanis, Clinical Evaluation of soft tissue esthetics around immediate implant using dual zone therapeutic concept versus buccal gap fill to bone level, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2508
Record Dates: First submitted 2018-12-03; First posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Immediate Implant and Bone Graft

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate implant with dual zone therapeutic concept (Experimental)
  Interventions: Procedure: dual zone concept
- immediate implant with buccal bone fill (Active Comparator)
  Interventions: Procedure: dual zone concept

INTERVENTIONS:
Procedure: dual zone concept — immediate implant with bone fill till soft tissue level

SUMMARY:
Immediate implant placement in the esthetic zone is very challenging procedure although it is documented as a promising procedure (Berglundh, Persson and Klinge, 2002)(Cosyn et al., 2011). Extraction is usually accompanied by remodeling of the hard tissues which is more crucial in the anterior maxilla as it affects soft tissue esthetics(Araujo and Lindhe, 2005)(Covani et al., 2004)(Juodzbalys and Wang, 2007). It is well established that implant placement without filling the buccal gap leads to noticeable amount of bone loss at the alveolar contour(Botticelli, Berglundh and Lindhe, 2004)(Sanz et al., 2010). The protocol of immediate implant and temporization serves to provide acceptable esthetic results but soft tissue stability around the implant restoration is not always satisfactory(Noelken et al., 2018).Amount of soft tissue recession can be specified following immediate implant placement, even with flapless technique there is a limited risk of midfacial recession(Cosyn, Hooghe and De Bruyn, 2012).It was found that inadequate bone grafting in the facial defect increases the chance of mid facial recession(Le, Borzabadi-Farahani and Pluemsakunthai, 2014).

DETAILED DESCRIPTION:
By definition, the dual zone can be divided into soft tissue zone and bone zone; the soft tissue zone is the vertical dimension change measured from the free gingival margin to the mid crest labially, the bone zone is the hard tissues measured from the crestal bone towards the apex(Chu et al., 2012). The concept of the dual zone aims to maintain the hard, soft tissue volume and the blood clot where the grafting material act as a scaffold containing them and this will enhance the initial healing compared to the classic protocol of bone filling till the buccal bone level(Chu et al., 2012). A recent study claims that the xenograft particles can be successfully incorporated within the soft tissue without inflammation enhancing the soft tissue profile(Araujo and Lindhe, 2005). The temporary restoration has shown socket sealing property which protect and contain the blood clot and the graft material enhancing healing,thus filling the gap without involvement of the soft tissue has been the rational for immediate implant placement(Trimpou G, Weigl P, Krebs M, 2010).The main benefit of the dual zone concept is maintaining the blood supply from the periosteum and endosteum producing maximum healing potential with preserving the soft tissue stability by filling the soft tissue zone with bone graft in addition to immediate temporization acting as socket seal(Chu et al., 2012).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have at least one non restorable tooth in the esthetic zone that needs to be extracted.
2. Patients with healthy systemic condition.(Brightman. 1994)
3. Patients aged from 20 to 45 years old.
4. Buccal bone thickness should be at least 1mm. (Morton et al., 2014)
5. Availability of bone apical and palatal to the socket to provide primary stability.(Morton et al., 2014)
6. Good oral hygiene.(Wiesner et al., 2010)
7. Accepts one year follow-up period (cooperative patients).
8. Patient provides an informed consent.
9. Adequate Inter-arch space for implant placement.
10. favorable occlusion (no traumatic occlusion)

Exclusion Criteria:

1. Patients with signs of acute infection related to the area of interest.
2. Patients with habits that may jeopardize the implant longevity and affect the results of the study such as parafunctional habits (Lobbezoo et al., 2006).
3. Current and former smokers (Lambert, Morris and Ochi, 2000)
4. Pregnant females.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-12-20 (Estimated); Primary Completion 2019-11-20 (Estimated); Study Completion 2020-11-20 (Estimated)

PRIMARY OUTCOMES:
Pink Esthetic Score | 12 months post surgery
  The PES is based on seven variables: mesial papilla, distal papilla, soft-tissue level, softtissuecontour, alveolar process deficiency,soft-tissue color and texture. Each variable shall be assessed with a 2-1-0 score,with 2 being the best and 0 being thepoorest score.The mesial and distal papilla will be evaluatedfor completeness, incompleteness orabsence. All other variables will be assessedby comparison to a reference tooth.(Fürhauser et al., 2005)

SECONDARY OUTCOMES:
Buccal bone thickness | 12 months post surgery
  using a specially designed device that will be screwed to the fixture. (Merheb et al., 2016)
Gingival Thickness | 12 months post surgery
  Will be measured using an anesthetic needle with a rubber stopper,transgingivally piercing tissues horizontally,perpendicular to the long axis of the tooth/implant until it contacts bone, at 9 different points; three readings: mesially, midbuccally and distally at three different levels; 2mm, 4mm and 6mm apical to the gingival margin.The lengthof the part of the instrument that penetratedinto the soft tissue is measured in mm.(Wiesner et al., 2010)
Keratinized tissue width | 12 months post surgery
  Will be measured by a periodontal probe from the gingival margin to the mucogingival junction, at the mid buccal area.
Post operative swelling | 12 months post surgery
  Verbal Rating Scale (VRS); absent(no swelling), slight (intraoral swelling at the operated area), moderate (moderate intraoral swelling at the operated area) and intense (intensive extraoral swelling extending beyond the operated area), assessed during the first 7 postoperative days. (García et al., 2008)
Post Surgical Patient Satisfaction: Questionnaire | 12 months post surgery
  A 3-item questionnaire is asked and the patients shall use a 7 point answer scale. (Kiyak et al., 1984)